CLINICAL TRIAL: NCT01718925
Title: Vitamin D, Fatigue and Patient Reported Outcome (PRO) in Chronic Somatic and Functional Disorders.
Brief Title: 25-hydroxyvitamin D and Fatigue: The VITALITY Study
Status: Completed | Type: Observational
Sponsor: Ostfold Hospital Trust (Other)
Collaborators: Karolinska Institutet (Other); Aarhus University Hospital (Other); Oslo University Hospital (Other); Alesund Hospital (Other); Helse Stavanger HF (Other Government); Sykehuset Telemark (Other Government); Sykehuset Innlandet HF (Other); Ostfold University College (Other)
Responsible Party: Sponsor
Other Study IDs: 3256
Record Dates: First submitted 2012-10-29; First posted 2012-11-01 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Irritable Bowel Syndrome; Inflammatory Bowel Disease; Diabetes; Rheumatoid Arthritis
MeSH Terms: conditions — Irritable Bowel Syndrome; Inflammatory Bowel Diseases; Diabetes Mellitus; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Inflammatory Bowel Disease: Ulcerative Colitis and Crohns's disease patients will be recruited from sqeduled outpatient follow-up
- Irritable Bowel Syndrome: Irritable Bowel patients will be recruited from sqeduled outpatient follow-up
- Rheumatoid Arthritis: Rheumatoid Arthritis patients will be recruited from sqeduled outpatient follow-up
- Diabetes Mellitus: Diabetes mellitus patients will be recruited from sqeduled outpatient follow-up

SUMMARY:
The burden of chronic disease is continuing to rise. Even though patients may be in remission or have quiescent disease, several studies have confirmed that symptoms, such as e.g., fatigue, is troublesome.

The primary aim of this study is to investigate whether or not there might be an association between levels of vitamin D and the subjective experience of fatigue in conditions, such as inflammatory bowel disease, diabetes mellitus, rheumatoid arthritis and irritable bowel syndrome.

Secondary aims is to study both the co-occurence and influence of pain, depression and anxiety.

DETAILED DESCRIPTION:
The burden of chronic disease is continuing to rise. Even though patients may be in remission or have quiescent disease, several studies have confirmed that symptoms, such as e.g., fatigue, is troublesome.Previous studies have confirmed that vitamin D deficiency is associated with both Crohn's disease and Rheumatoid Arthritis. Since Vitamin D is associated with both onset of chronic disease and energy, we aim in this study to assess its impact on fatigue in various chronic diseases.

The primary aim of this study is to investigate whether or not there might be an association between levels of vitamin D and the subjective experience of fatigue in conditions, such as inflammatory bowel disease, diabetes mellitus, rheumatoid arthritis and irritable bowel syndrome.

Secondary aims is to study both the co-occurence and influence of pain, depression and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* informed consent,
* over 18 years of age

Exclusion Criteria:

* dementia,
* cognitive disorders,
* not able to comply with the study procedures,
* on active vitamin D treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an established diagnose of IBD, DIA, IBS or RA is eligible for inclusion in this study. Patients must be over 18 years of age. Disease activity will be measured using the SCCAI for ulcerative colitis, SCDAI for Crohn's disease, DAS-28 for rheumatoid arthritis. In Dia and IBD objective activity measures, such as calprotectin in stools and HbA1C, will be collected.
Sampling Method: Non-Probability Sample
Enrollment: 614 (Actual)
Dates: Start 2012-10; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Fatigue | 2 years
  Fatigue and the impact of vitamin d levels

CONTACTS AND LOCATIONS:
Overall Officials: Lars-Petter Jelsness-Jørgensen, PhD, Principal Investigator — Ostfold Hospital Trust